CLINICAL TRIAL: NCT00181090
Title: Use of the Atkins Diet for Children With Intractable Epilepsy: A Comparison of Daily Carbohydrate Limits
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-01-26-05
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Ketosis; Atkins; seizures
MeSH Terms: conditions — Epilepsy; Ketosis; Seizures

INTERVENTIONS:
Behavioral: Modified Atkins diet

SUMMARY:
This study is designed to further investigate the use of a modified Atkins diet for children with intractable, daily seizures. It is a follow-up to a study recently completed by our institution. In this 6-month study, children will be randomized to either 10 or 20 grams of carbohydrate per day, then crossed over to the opposite amount at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-18
* Daily seizures or 7 per week
* Failed at least 2 anticonvulsants

Exclusion Criteria:

* Prior use of the Atkins diet for over 1 week
* Significant heart, liver, or kidney disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2005-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Seizure control | 6 months
Ketosis | 6 months

SECONDARY OUTCOMES:
Tolerability | 6 months
Safety - cholesterol, kidney function, weight | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, Krauss GL, McGrogan JR, Freeman JM. Efficacy of the Atkins diet as therapy for intractable epilepsy. Neurology. 2003 Dec 23;61(12):1789-91. doi: 10.1212/01.wnl.0000098889.35155.72. PMID 14694049
- See also: Family and patient created website for study patients — http://www.atkinsforseizures.com